CLINICAL TRIAL: NCT04713735
Title: A Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Impact of Lactoferrin Dietary Supplementation on Respiratory Tract Infections in an Elderly Population
Brief Title: Impact of Lactoferrin, a Dietary Supplement, vs. Placebo on Respiratory Tract Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 3393-1
Record Dates: First submitted 2021-01-08; First posted 2021-01-19 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-03

CONDITIONS: Immune Health

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Placebo (Placebo Comparator): Control: Placebo
  Interventions: Dietary Supplement: Control: Placebo
- Investigational: 600 mg bovine lactoferrin supplement (Experimental): Investigational: 600 mg bovine lactoferrin supplement
  Interventions: Dietary Supplement: bovine lactoferrin supplement

INTERVENTIONS:
Dietary Supplement: Control: Placebo — Placebo
  Arms: Control: Placebo
Dietary Supplement: bovine lactoferrin supplement — 600 mg
  Arms: Investigational: 600 mg bovine lactoferrin supplement

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate the impact of bovine Lactoferrin (bLf) on respiratory tract infections (RTIs) in an elderly population in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 55 years of age at time of consent
* Able to eat and drink, with assistance if required
* Investigator and Community Living Center administration expect subject to reside in Community Living Center for the duration of the study
* Signed consent obtained from subject or legally authorized representative
* Signed authorization obtained to use and/or disclose Protected Health Information

Exclusion Criteria:

* Receiving (or, in the opinion of the Investigator, likely to receive in the next 6 months) parenteral nutrition
* Have a known eating disorder or illness, which requires a therapeutic diet incompatible with fortification and/or supplementation
* Has been diagnosed as immunocompromised or is receiving medication which may cause immune compromise. Note relative immunocompromisation due to age would not exclude the subject
* Known allergy or intolerance to study products
* On an end-of-life care pathway or, in the opinion of the Investigator, has a life expectancy of less than 6 months
* Inappropriate for inclusion in the study in the opinion of the Investigator or Community Living Center administration
* Have experienced Respiratory Tract Infection within 1 week prior to randomization

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Number of Respiratory Tract Infections | 365 days

SECONDARY OUTCOMES:
Severity of Respiratory Tract Infection | 365 days
  Mild, Moderate, or Severe rating
Duration of Respiratory Tract Infection | 365 days
Number of Respiratory Tract Infections | 180 days
Treatment of Respiratory Tract Infections | 365 days
Complications from Respiratory Tract Infections | 365 days
Microorganism causing Respiratory Tract Infection | 365 days
Level of protective antibody against influenza virus | Baseline, Day 45, Day 90, Day 180, Day 270, and Day 365
Inflammatory cytokine | Baseline, Day 45, Day 90, Day 180, Day 270, and Day 365
Protection against apoptosis and oxidative stress | Baseline, Day 45, Day 90, Day 180, Day 270, and Day 365
Salivary level of lactoferrin | Baseline, Day 45, Day 90, Day 180, Day 270, and Day 365
Salivary level of thiocyanate | Baseline, Day 45, Day 90, Day 180, Day 270, and Day 365
Salivary level of hypohalous acid | Baseline, Day 45, Day 90, Day 180, Day 270, and Day 365
Complete Blood Count | Baseline, Day 45, Day 90, Day 180, and Day 365
Comprehensive Metabolic Panel | Baseline, Day 45, Day 90, Day 180, and Day 365
Body Weight | Baseline, Day 45, Day 90, Day 180, and Day 365
Short Form (12) Health Survey Version 2 (SF-12v2®) | Baseline, Day 45, Day 90, Day 180, and Day 365
Use of medical treatments | 365 days
Medically confirmed Adverse Events | 365 days
COVID Vaccine specific inflammatory panel | Day 45, Day 90, Day 180, Day 270, and Day 365
  IGG concentrations and geometric means of SARS psuedovirus neutralization titers and Cytokines
Influenza Hemagglutination-inhibition Antibody Titer | Pre-booster, Post-booster day 2, Post-booster day 7, and Post-booster day 28
Cytokine Panel | Pre-booster, Post-booster day 2, Post-booster day 7, and Post-booster day 28

CONTACTS AND LOCATIONS:
Overall Officials: Steven Wu, MD, Study Director — Mead Johnson/RB
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No